CLINICAL TRIAL: NCT04503460
Title: Mechanisms of Adverse Effects of Long-Acting Beta-Agonists in Asthma
Acronym: MAELABA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: European Research Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 19SM5101; 2019-003036-23 (EudraCT Number)
Record Dates: First submitted 2019-07-01; First posted 2020-08-07 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Asthma
Keywords: Asthma; Salmeterol; Fluticasone
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Intervention Model Description: All participants will receive salmeterol xinafoate monotherapy for 2 weeks, followed by a washout period for 2 weeks, followed by salmeterol xinafoate/fluticasone propionate combination therapy for 2 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single treatment arm (Experimental): All participants who are deemed eligible for inclusion in the study following screening will be enrolled into a single experimental arm which will comprise the following sequential stages:
  1. Baseline sampling; participants only use 'as required' ipratropium bromide when needed (1 week)
  2. Salmeterol xinafoate monotherapy 50 μg twice in the morning and twice in the evening + 'as required' ipratropium bromide when needed (2 weeks)
  3. Washout period; participants only use 'as required' ipratropium bromide when needed (2 weeks)
  4. Salmeterol xinafoate 50 μg / fluticasone propionate 250 μg combination therapy twice in the morning and twice in the evening + 'as required' ipratropium bromide when needed (2 weeks)
  Interventions: Drug: Salmeterol Xinafoate; Drug: Salmeterol Fluticasone

INTERVENTIONS:
Drug: Salmeterol Xinafoate — All participants will receive inhaled salmeterol xinafoate 50 μg twice in the morning and twice in the evening for 2 weeks; this will be followed by a 2-week washout period during which time no beta-agonists will be administered. Participants will be asked to use 'as required' ipratropium bromide during this period when needed in place of short-acting beta agonists.
Drug: Salmeterol Fluticasone — Following the 2-week washout period, all participants will receive inhaled salmeterol xinafoate 50 μg combined with fluticasone propionate 250 μg twice in the morning and twice in the evening for 2 weeks. Participants will be asked to use 'as required' ipratropium bromide during this period when needed in place of short-acting beta agonists.

SUMMARY:
This study aims to elucidate the pathophysiological mechanisms underlying the adverse effects associated with the use of long-acting beta-agonists (LABAs) in asthma. Participants with mild asthma will be enrolled into a single-arm, unblinded trial in which they receive 2 weeks of salmeterol xinafoate monotherapy, followed by a 2-week washout period, followed by 2 weeks of salmeterol xinafoate / fluticasone propionate combination therapy. The induction of asthma disease-relevant pro-inflammatory mediators in the airways will be measured at each stage and correlated with relevant clinical parameters.

DETAILED DESCRIPTION:
The use of long-acting beta-agonists (LABAs) alone to treat asthma has been associated with increased mortality rates. Between 2012 and 2013, 3% of patients who died from asthma in the UK were found to be on LABA monotherapy, despite guidelines recommending that LABAs must always be administered with inhaled corticosteroids (ICS). Monotherapy with the LABA salmeterol has been linked to a significant increase in asthma-related mortality rates when used without ICS. When salmeterol is used with ICS, it is not associated with an increased risk of serious asthma-related events and is associated with fewer exacerbations than when using ICS alone. The purpose of this study is to understand the mechanisms underlying why LABA use on its own causes worse outcomes in asthma patients. If the mechanisms can be successfully understood, this could provide further compelling evidence to optimise safe of these medicines in airway disease.

The primary objective of this study will be: to determine whether LABA monotherapy with salmeterol for 2 weeks in asthmatic patients induces disease-relevant mediators (as identified through ex vivo studies) in the airways in vivo; and to determine whether LABA/ICS combination therapy with salmeterol xinafoate/fluticasone propionate for 2 weeks in the same asthmatic patients will abolish the induction of disease-relevant mediators in the airways in vivo. If it can be shown that the levels of these inflammatory mediators increase in the airways of asthmatic patients when they are on salmeterol xinafoate monotherapy, and that this effect is decreased when asthmatic patients are on salmeterol xinafoate /fluticasone propionate combination therapy, this will provide evidence for a mechanism underlying the adverse effects of salmeterol in asthmatic patients.

Secondary objectives will be to determine the impact of LABA monotherapy with salmeterol xinafoate for 2 weeks and LABA/ICS therapy with salmeterol xinafoate/fluticasone propionate for 2 weeks on the following parameters in asthmatic patients: lung function (assessed by spirometry); airway inflammation (assessed by measuring fractional exhaled nitric oxide); airway hyperresponsiveness (assessed by histamine challenge testing); asthma symptom control (assessed by the Asthma Control Questionnaire-6); and serum brain-derived neurotrophic factor (BDNF) concentration and platelet BDNF concentration.

ELIGIBILITY:
INCLUSION CRITERIA

* Age > 18 years
* A doctor's diagnosis of asthma (mild in severity)
* No current regular asthma treatment or regular asthma treatment in the preceding 6 weeks; only a history of using short-acting bronchodilator inhalers on demand is allowed
* Pre-bronchodilator FEV1 value > 70% of the predicted value

EXCLUSION CRITERIA

* History or evidence of chronic respiratory disease other than asthma
* History or evidence of other disease, blood test results outside the normal reference range or medication use that would impair the ability of participants to safely undertake the study or the ability of researchers to interpret the study results; this includes, but is not limited to, the use of anticoagulants (e.g. warfarin), adenosine diphosphate (ADP) receptor inhibitors (e.g. clopidogrel), antiretroviral therapy (due to the potential for interaction with fluticasone), certain antifungal agents (due to the potential for interaction with fluticasone) and beta-blockers
* Current use or use in the last 6 weeks of systemic or nasal topical steroids, inhaled corticosteroids or systemic immunosuppressants
* Platelet count < 150 x 109/L or international normalised ratio (INR) > 1.5
* History of smoking > 5 pack years, current smoker or history of smoking in the last 4 weeks
* Current vaping or history of vaping in the last 4 weeks
* Current illicit drug use/abuse
* Abnormal chest x-ray appearance
* Signs or symptoms of upper respiratory tract infection or lower respiratory tract infection in the preceding 6 weeks
* Cardiac conduction abnormalities on electrocardiogram (ECG)
* Current pregnancy or planning to become pregnant during the study period
* Breastfeeding during the study period
* Inability to provide informed consent to participate in the study
* Current involvement in any other clinical research studies involving medicinal products or devices; or involvement in clinical research studies involving medicinal products within the last 30 days or within 5 half-lives of the medicinal product (whichever is longer)
* Inability to speak English or inability to understand verbal or written English
* Inability to attend hospital for all scheduled study visits
* Hypersensitivity to any of the investigational medicinal products (IMPs) or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
1. Pro-inflammatory mediator protein expression following salmeterol monotherapy | [Time Frame: Change between Day 1 (baseline bronchoscopy) and Day 15 (post-salmeterol monotherapy bronchoscopy)]
  Change from baseline in the level of disease-relevant pro-inflammatory mediator IL-6 in Bronchoalveolar Lavage (BAL) fluid following 2 weeks of salmeterol monotherapy.

OTHER OUTCOMES:
1. Pro-inflammatory mediator gene expression following salmeterol monotherapy | [Time Frame: Change between Day 1 (baseline bronchoscopy) and Day 15 (post-salmeterol monotherapy bronchoscopy)]
  Change from baseline in the levels of gene expression of disease-relevant pro-inflammatory mediators in BAL fluid following 2 weeks of salmeterol monotherapy.
2. Pro-inflammatory mediator protein expression following salmeterol/fluticasone combination therapy | [Time Frame: Change between Day 29 (post-salmeterol washout bronchoscopy) and Day 43 (post salmeterol/fluticasone combination therapy bronchoscopy)]
  Change from baseline in protein levels of disease-relevant pro-inflammatory mediators in BAL fluid following 2 weeks of salmeterol/fluticasone combination therapy
3. Pro-inflammatory mediator gene expression following salmeterol/fluticasone combination therapy | [Time Frame: Change between Day 29 (post-salmeterol washout bronchoscopy) and Day 43 (post salmeterol/fluticasone combination therapy bronchoscopy)]
  Change from baseline in the levels of gene expression of disease-relevant pro-inflammatory mediators in BAL fluid following 2 weeks of salmeterol/fluticasone combination therapy
4. Lung function (spirometry) | [Time Frame: Over 7 weeks]
  Change in lung function, measured by spirometry, between baseline and following 2 weeks of salmeterol monotherapy; and between post-salmeterol washout baseline and following 2 weeks salmeterol/fluticasone combination therapy
5. Fractional exhaled nitric oxide | [Time Frame: Over 7 weeks]
  Change in fractional exhaled nitric oxide between baseline and following 2 weeks of salmeterol monotherapy; and between post-salmeterol washout baseline and following 2 weeks salmeterol/fluticasone combination therapy
6. Airway hyperresponsiveness (histamine challenge) | [Time Frame: Over 7 weeks]
  Change in airway hyperresponsiveness, measured by histamine challenge, between baseline and following 2 weeks of salmeterol monotherapy; and between post-salmeterol washout baseline and following 2 weeks salmeterol/fluticasone combination therapy
7. Asthma symptom control (Asthma Control Questionnaire 6 / ACQ-6 score) | [Time Frame: Over 7 weeks]
  Change in asthma symptom control, measured by ACQ-6 scoring, between baseline and following 2 weeks of salmeterol monotherapy; and between post-salmeterol washout baseline and following 2 weeks salmeterol/fluticasone combination therapy. ACQ-6 is a validated tool for assessing patients' perceived degree of severity and symptom control of their asthma. The questionnaire comprises of 6 multiple choice questions, each with 7 possible choices (only one selectable) carrying scores between 0 and 6 - total added ACQ-6 score ranges between 0 and 36, with a score of 36 representing the highest possible symptom burden measured by this questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian L Johnston, MBBS PhD FRCP FRSB FMedSci, Study Chair — Imperial College London
Locations (1):
- St Mary's Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study data to be stored in an online repository for potential future sharing with other researchers. Current protocol and other related documents are undergoing amendments in order to include this plan.